CLINICAL TRIAL: NCT00773513
Title: A Randomized, Controlled, Open-Label, Multi-Centre, Parallel-Group Study To Assess All-Cause Mortality And Cardiovascular Morbidity In Patients With Chronic Kidney Disease On Dialysis And Those Not On Renal Replacement Therapy Under Treatment With MIRCERA® Or Reference ESAs.
Brief Title: A Study to Assess All-Cause Mortality and Cardiovascular Morbidity in Participants With Chronic Kidney Disease (CKD) on Dialysis and Those Not on Renal Replacement Therapy Receiving Methoxy Polyethylene Glycol-Epoetin Beta (Mircera) or Reference Erythropoietin Stimulating Agents (ESAs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH21260; 2007-005129-31
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chronic Renal Anemia
MeSH Terms: interventions — Darbepoetin alfa; Epoetin Alfa; epoetin beta; continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erythropoiesis Stimulating Agents (Active Comparator): Participants will receive reference ESA according to approved label. The approved reference ESA compounds in the study will be darbepoetin alfa, epoetin alfa and epoetin beta.
  Interventions: Drug: Darbepoetin Alfa; Drug: Epoetin Alfa; Drug: Epoetin Beta; Drug: methoxy polyethylene glycol-epoetin beta
- Methoxy Polyethylene Glycol-Epoetin Beta (Experimental): Participants not currently being treated with an ESA will receive methoxy polyethylene glycol-epoetin beta iv or sc once every 2 weeks for correction of renal anemia (target Hb 10-12 g/dL). Once corrected and in participants currently being treated with an ESA, methoxy polyethylene glycol-epoetin beta will be administered once monthly.
  Interventions: Drug: Darbepoetin Alfa; Drug: Epoetin Alfa; Drug: methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Darbepoetin Alfa — Darbepoetin alfa will be administered as per approved label.
  Other Names: Aranesp®, Nespo®, Aranest®
Drug: Epoetin Alfa — Epoetin alfa will be administered as per approved label.
  Other Names: Eprex®, Epogen®, Epopen®, Erypo®
Drug: Epoetin Beta — Epoetin beta will be administered as per approved label.
  Other Names: Neorecormon®, Recormon®
  Arms: Erythropoiesis Stimulating Agents
Drug: methoxy polyethylene glycol-epoetin beta — Participants who are currently not being treated with an ESA will receive methoxy polyethylene glycol-epoetin beta administered at a starting dose of 0.6 mcg/kg body weight once every 2 weeks. Participants who are currently being treated with an ESA will receive methoxy polyethylene glycol-epoetin beta at a dose of 120, 200 or 360 mcg once monthly (based on ESA dose administered in Week -1)
  Other Names: Mircera®

SUMMARY:
This 2 arm safety study will compare the outcome with respect to a composite endpoint of all-cause mortality and non-fatal cardiovascular events (myocardial infarction, stroke) in CKD participants either on dialysis or not receiving renal replacement therapy under treatment with methoxy polyethylene glycol-epoetin beta or reference ESAs. Participants will be randomized to receive intravenous (iv) or subcutaneous (sc) methoxy polyethylene glycol-epoetin beta at the following doses: for participants not already receiving ESA treatment, methoxy polyethylene glycol-epoetin beta will be administered at a starting dose of 0.6 micrograms per kilograms every 2 weeks (mcg/kg/2wks) iv or sc; for participants receiving maintenance ESA treatment, iv or sc methoxy polyethylene glycol-epoetin beta will be administered at an initial monthly dose of 120, 200 or 360 micrograms (mcg) depending on the weekly dose of ESA received prior to first methoxy polyethylene glycol-epoetin beta administration. Participants randomized to reference ESA treatment will receive iv or sc ESAs in accordance with their prescribed dosing information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with symptomatic anemia associated with CKD
* Participants with renal anemia who are not treated with an ESA:
* Anemia was defined as hemoglobin (Hb) concentration less than (<) 11.0 grams per deciliter (g/dL) (mean of 2 screening values with at least one day and a maximum of 2 weeks between measurements) with clinical indication for ESA treatment
* Participants with renal anemia who are on maintenance ESA therapy:
* If on dialysis: regular long-term hemodialysis or peritoneal dialysis therapy with the same mode of dialysis for at least 3 months before screening
* Hb concentration between 10 and 12 g/dL (mean of 2 screening values with at least one day and a maximum of 2 weeks between measurements)
* Participants with adequate iron status defined as: serum ferritin above or equal to 100 micrograms per liter or transferrin saturation above or equal to 20 percent

Exclusion Criteria:

* Contraindications to ESA treatment: uncontrolled hypertension, hypersensitivity to the active substance or any of the excipients, any other contraindication to ESA therapy
* Conditions known to cause inadequate response to ESA treatment or anemia other than symptomatic anemia associated with CKD:
* History of hemoglobinopathy
* Anemia due to hemolysis
* Pure red cell aplasia
* High likelihood of early withdrawal (for example, within 1 year) or interruption of the study
* Pregnancy or breast-feeding
* Women of childbearing potential without effective contraception
* Administration of another investigational drug within 1 month before screening or planned during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2825 (Actual)
Dates: Start 2008-12-12 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (196):
- Argentina (4):
  - Fresenius Medical Care Martinez, Buenos Aires
  - Fresenius Medical Care Morón, Buenos Aires
  - Fresenius Medical Care San Martin, Buenos Aires
  - Fresenuis Medical Care Mansilla, CABA
- Australia (8):
  - Gosford Hospital; Renal, Gosford, New South Wales
  - Renal Research Dr Simon Roger, Gosford, New South Wales
  - Cairns Hospital; Renal Services, Cairns, Queensland
  - Gold Coast Hospital Department of Pharmacology & Therapeutics, Southport, Queensland
  - ROYAL ADELAIDE HOSPITAL; Renal Clinical Trials, CNARTS, Adelaide, South Australia
  - Launceston General Hospital; Diabetes and Renal Research Unit, Launceston, Tasmania
  - Monash Medical Centre; Renal Transplant Unit, Clayton, Victoria
  - Royal Perth Hospital; Nephrology, Perth, Western Australia
- Belgium (5):
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - AZ Delta (Campus Wilgenstraat), Roeselare
- Brazil (10):
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - PUCPR, Curitiba, Paraná
  - Hospital Univ. Pedro Ernesto - Hupe; Nefrologia, Rio de Janeiro, Rio de Janeiro
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo, São Paulo
  - Clinica de Medicina Interna e Nefrologia (CMIN), São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP; Nefrologia, São Paulo, São Paulo
  - Instituto de Hemodialise Sorocaba, Sorocaba, São Paulo
- Croatia (7):
  - General Hospital Karlovac; Dept of Haemodialysis, Karlovac
  - Clinical Hospital Osijek; Dept of Haemodialysis, Osijek
  - Clinical Hospital Center Rijeka; Dialysis, Rijeka
  - General Hospital Josip Bencevic; Department of Haemodialysis, Slavonski Brod
  - Clinical Hospital Split; Dialysis, Split
  - General Hospital Zadar; Dialysis, Zadar
  - Klinicki Bolnicki Centar Zagreb; Dialysis, Zagreb
- Czechia (4):
  - Fakultni Nemocnice Kralovske Vinohrady (FNKV); Interni Hematologicka Klinika, Hradec Králové
  - Faculty Hospital; Dialysis Unit, Ostrava
  - Institut Klinicke A Experimentalni Mediciny Klinika Nefrologie, Prague
  - Nemocnice Strahov; Interni Oddeleni-Strahov, Prague
- France (18):
  - Centre Hospitalier; Hemodialyse, Annonay
  - Hopital Pellegrin; Departement Nephrologie, Bordeaux
  - Centre Hospitalier Du Dr Duchenes; Service De Nephrologie & Hemodialyse, Boulogne
  - Hopital La Cavale Blanche; Nephrologie, Brest
  - Hopital Louis Pasteur; Nephrologie - Hemodialyse, Colmar
  - Clinique Lambert; Service de Néphrologie dialyse, La Garenne-Colombes
  - Chu Dupuytren; Nephrologie-Hemodialyse, Limoges
  - Aural, Lyon
  - Hopital Edouard-Herriot; Nephrologie - Hemodialyse, Lyon
  - Centre Hospitalier Les Chanaux; Service de Néphrologie Unité 12, Mâcon
  - Service de Nephrologie & D'Immunologie; Clinique, Nantes
  - Centre Hospitalier Uni Ire Gaston Doumergue; Service D'Hemodialyse, Nîmes
  - Aura - Centre Henri Kunt Ziger, Paris
  - Hopital Laennec; Echo, Saint-Herblain
  - Hopital Sud ; Nephrologie Hemodialyse, Salouël
  - Hopital Civil; Nephrologie Clinique Medicale B, Strasbourg
  - Hopital Rangueil; Nephrologie Hemodialyse, Toulouse
  - Ch De Valenciennes; Nephrologie, Valenciennes
- Germany (18):
  - Gemeinschaftspraxis Dr. Stefan Zinn und Steffen Hengst, Alsfeld
  - KFH Nierenzentrum Bad Hersfeld; Nephrologie, Bad Hersfeld
  - Universitätsklinikum Bonn; Medizinische Klinik und Poliklinik I; Allgemeine Innere Medizin, Bonn
  - Dialysepraxis Dr. med. Uwe Kraatz, Demmin
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf
  - Universitätsklinikum Duesseldorf; Klinik fuer Nephrologie, Düsseldorf
  - Universitätsklinikum Erlangen; Medizinische Klinik 4; Nephrologie und Hypertensiologie, Erlangen
  - Georg-Haas-Dialysezentrum der PHV, Giessen
  - Nephrologische Schwerpunktpraxis; Hamburg Barmbek, Hamburg
  - Klinikum Hann. Münden, Nephrologisches Zentrum Niedersachsen, Hannoversch Münden
  - Uniklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes; Klinik f. Innere Medizin IV, Homburg/Saar
  - UNI-Klinikum Campus Kiel Klinik f.Innere Medizin IV, Kiel
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V.; KfH-Nierenzentrum, München
  - KFH Nierenzentrum Oberschleissheim, Oberschleißheim
  - Dres. Roland Erwin Winkler Ann Michelsen Dietmar Sehland u.w., Rostock
  - Praxis Dr.med. Joachim Leicht, Schwandorf in Bayern
  - Robert-Bosch-Krankenhaus; Allgemeine Innere Medizin und Nephrologie, Stuttgart
- Greece (5):
  - Uni Hospital of Alexandroupoli; Nephrology Dept., Alexandroupoli
  - Laiko General Hospital; Nephrology Div., Athens
  - Uni Hospital of Ioannina; Nephrology Dept., Ioannina
  - Univeristy Hospital of Larissa; Nephrology, Larissa
  - Hippokratio Hospital; Nefrology, Thessaloniki
- Israel (5):
  - Rabin MC- Belinson campus, Petah Tikva
  - Rabin MC- Hasharon campus, Petah Tikva
  - Sheba MC; Nephrology, Ramat Gan
  - Sourasky MC; Dept. of Nephrology, Tel Aviv
  - Assaf-Harofeh MC; Nephrology, Zrifin
- Italy (28):
  - Ospedale Bernardo Ramazzi; U.O. Di Nefrologia E Dialisi, Carpi, Emilia-Romagna
  - Ospedale Civile; Servizio Di Nefrologia E Dialisi, Imola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Nefrologia E Dialisi, Modena, Emilia-Romagna
  - Ospedale Maggiore; U.O.Complessa di Nefrologia e Dialisi, Parma, Emilia-Romagna
  - Ospedale Civile; Divisione de Nefrologia E Dialisi, Piacenza, Emilia-Romagna
  - Ospedale Provinciale S. Maria delle Croci; Divisione Nefrologia e Dialsi, Ravenna, Emilia-Romagna
  - A.O. Santa Maria Nuova Di Reggio Emilia; Unita Operativa Di Nefrologia E Dialisi, Reggio Emilia, Emilia-Romagna
  - Universita' Di Tor Vergata; Clinica Nefrologia Dialisi, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova; Nefrologia, Genoa, Liguria
  - Ospedale Caduti Bollatesi; U.O. Nefrologia E Dialisi, Bollate, Lombardy
  - ASST DI LECCO; Nefrologia e Dialisi, Lecco, Lombardy
  - Presidio Ospedaliero Maggiore Policlinico Fondazione IRCCS; Pad Croff Div Nefrologia Dialisi, Milan, Lombardy
  - ASST SANTI PAOLO E CARLO; U.O.S. Nefrologia e Dialisi, Milan, Lombardy
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA; Dipartimento di Nefrologia e Dialisi, Milan, Lombardy
  - Fondazione Salvatore Maugeri; Divisione Di Nefrologia E Dialisi, Pavia, Lombardy
  - ASST LARIANA; Divisione di Nefrologia e Dialisi, S Fermo Della Battaglia, Lombardy
  - Ospedale S. Marta S. Venera Nuovo; U.O. Nefrologia Dialisi, Acireale, Sicily
  - Azienda Ospedaliera Cannizzaro Unità Operativa Nefrologia, Catania, Sicily
  - A.O.U. Policlinico G.Martino; U.O.C. Nefrologia e Dialisi, Messina, Sicily
  - Azienda Ospedaliera San Salvatore; Divisione Nefrologia E Dialisi, Pesaro, The Marches
  - Presidio Ospedaliero Di Lodi; U.O. Nefrologia E Dialisi, LODI, Tuscany
  - Nuovo Ospedale Di Prato, Prato, Tuscany
  - Ospedale S. Giacomo; U.O. Di Nefrologia e Dialisi, Castelfranco, Veneto
  - Azienda Ospedaliera Sant'Anna Unità Operativa Complessa di Nefrologia Dialisi, Cona (FE), Veneto
  - P.O. Di Conegliano; U.O. Di Nefrologia E Dialisi, Conegliano, Veneto
  - Az. Osp. Di Padova; U.O. Nefrologia 2 E Dialisi, Padua, Veneto
  - Azienda Ospedaliera Santa Maria Misericordia; Divisione Nefrologia Dialisi, Rovigo, Veneto
  - A.O. Cà Foncello; U.O.Nefrologia, Dialisi e Centro Trapianti, Treviso, Veneto
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinic, Nephrology Center, Vilnius
- Malaysia (3):
  - University Malaya Medical Centre; Division of Nephrology, Department of Medicine, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Hospital Kuala Lumpur; Department of Medicine, Kuala Lumpur
  - Selayang Hospital; Dept of Medicine, Kuala Selangor
- Investigación Nefrológica S.C., Cuernavaca, Morelos, Mexico
- Centro Especializado San Fernando; Nefrología, Diálisis y Trasplante Renal, Panama City, Panama
- Philippines (2):
  - Cebu Doctors University Hospital, Cebu City
  - National Kidney and Transplant Institute, Quezon City
- Poland (14):
  - Akademia Medyczna; Klinika Nefrologii I Chorob Wewnetrznych, Bydgoszcz
  - Specjalistyczny Szpital Wojewodzki w Ciechanowie; Oddzial Nefrologiczny, Ciechanów
  - Fresenius Nephrocare Polska Sp zo.o.Centrum Dializ Fresenius Osrodek Dializ Nr 45 w Dabrowie Tarn, Dąbrowa Tarnowska
  - NZOZ Stacja Dializ Hand-Prod w Gorlicach, Gorlice
  - Fresenius Nephrocare Polska Sp zo.o. Centrum Dializ Fresenius Osrodek Dializ Nr 42 w Jasle, Jasło
  - NZOZ Stacja Dializ Hand-Prod w Limanowej, Limanowa
  - Fresenius Nephrocare Polska Sp. z o.o., Centrum Dializ Fresenius, Osrodek Dializ nr 53 w Pabianicach, Pabianice
  - Fresenius Nephrocare Polska Sp. z o.o., Centrum Dializ Fresenius, Osrodek Dializ numer 71 w Poznaniu, Poznan
  - Stacja Dializ NZOZ Centrum Medyczne MEDYK, Rzeszów
  - Fresenius Nephrocare Polska Sp.zo.o.Centrum Dializ FreseniusOśrodek Dializ Nr 62 w Sandomierzu, Sandomierz
  - Wojewodzki Szpital Zespolony, Stacja Dializ, Skierniewice, Skierniewice
  - Powiatowy Szpital Specjalistyczny w Stalowej Woli; Oddział Nefrologii i Dializoterapii, Stalowa Wola
  - Specjalistyczny Szpital im A.Sokołowskiego w Wałbrzychu; Oddzial Nefrologiczny, Wałbrzych
  - S.P. Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
- Russia (4):
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg, Sankt-Peterburg
  - St.Petersburg State Budget Institution of Healthcare "City Mariinskaya Hospital", Saint Petersburg
  - SBEI of HPE "Northwestern State Medical University n.a. I.I.Mechnikov" of MoH of RF, Saint Petersburg
  - St.Petersburg State Budget Institution of Healthcare "City Hospital Saint Hosiomartyr Elisabeth"., Saint Petersburg
- Serbia (5):
  - Clinical Center of Serbia; Clinic of Urology, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Zemun Hospital; Nephrology, Belgrade
  - Clinical Center Nis; Clinic for Nephrology and Hemodialysis, Niš
  - Clinical Center Voivodina; Clinic for Immunology and Nephrology, Novi Sad
- Singapore (3):
  - National University Hospital; Dept of Medicine, Singapore
  - Singapore General Hospital; Renal Medicine, Singapore
  - Tan Tock Seng Hospital; Department of Renal Medicine, Singapore
- South Korea (2):
  - Seoul National Uni Hospital; Internal Medicine, Seoul
  - Samsung Medical Center; Nephrology Department, Seoul
- Spain (13):
  - Hospital Txagorritxu; Servicio de Nefrologia, Vitoria-Gasteiz, Alava
  - Complejo Hospitalario Torrecardenas; Servicio de Nefrologia, Almería, Almeria
  - Hospital Severo Ochoa; Servicio de Nefrologia, Leganés, Madrid
  - Hospital Infanta Sofia; Servico de Nefrologia, San Sebastián de los Reyes, Madrid
  - Hospital de Navarra; Servicio de Nefrologia, Pamplona, Navarre
  - Hospital de Cruces; Servicio de Nefrologia, Barakaldo, Vizcaya
  - Hospital de Basurto; Servicio de Nefrologia, Bilbao, Vizcaya
  - Hospital de Galdakano; Servicio de Nefrologia, Galdakao, Vizcaya
  - Hospital del Mar; Servicio de Nefrologia, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Complejo Hospitalario de Jaen- Hospital Universitario Medico Quirurgico, Jaén
  - Hospital Ramon y Cajal; Servicio de Nefrologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Nefrologia, Madrid
- Sweden (3):
  - Danderyds Sjukhus; Dept. of Nephrology, Danderyd
  - Maelar Hospital; Department of Medicine, Eskilstuna
  - Uppsala University Hospital; Department of Internal Medicine, Nephrology Section, Uppsala
- Taiwan (2):
  - Chang Gung Medical Fundation Kaohsiung Branch; Nephrology, Kaohsiung City
  - National Taiwan Uni Hospital; Nephrology Dept, Taipei
- Thailand (3):
  - King Chulalongkorn Memorial Hospital; Renal Unit, Department of Medicine, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Dept. of Medicine, Renal Division, Chiang Mai
  - Buddhachinaraj Hospital Renal Division; Dept of Medicine, Phitsanulok
- Turkey (Türkiye) (3):
  - Cukurova University School of Medicine; Nefrology Department, Adana
  - Baskent University Hospital; Transplantation, Ankara
  - Inonu Uni School of Medicine, Malatya
- United Kingdom (23):
  - Ulster Hospital; Nephrology, Belfast
  - Belfast City Hospital; Nephrology Unit, Belfast
  - St Luke'S Hospital; Renal Unit, Bradford
  - University Hospital of Wales; Institute of Nephrology, Cardiff
  - St Helier Hospital; Renal Unit, Carshalton
  - University Hospital Coventry And Warwickshire Nhs Trust; Department Of Nephrology, Coventry
  - Dorset County Hospital; Renal Unit, Dorchester
  - Royal Devon & Exeter Hospital; Dept of Nephrology, Exeter
  - Hull Royal Infirmary; Renal Medicine, Hull
  - The Ipswich Hospital Nhs Trust; The Renal Unit, Ipswich
  - St James Uni Hospital; Renal Unit, Leeds
  - Leicester General Hospital; Dept of Nephrology, Leicester
  - Royal Free & University College Medical School; Centre for Nephrology, London
  - James Cook Hospital; Nephrology, Middlesbrough
  - Freeman Hospital; Nephrology, Newcastle upon Tyne
  - The Churchill; Oxford Kidney Unit, Oxford
  - Derriford Hospital; Department Of Renal Medicine, Plymouth
  - Royal Preston Hospital; Department of Renal Medicine, Preston
  - Salford Royal Foundation Trust; Department Of Nephrology, Salford
  - Royal Shrewsbury Hospital, Shrewsbury
  - Morriston Hospital; Renal Medicine, Swansea
  - Royal Cornwall Hospital; Renal Unit, Truro
  - Worthing Hospital; Renal Unit, West Sussex

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Locatelli F, Hannedouche T, Fishbane S, Morgan Z, Oguey D, White WB. Cardiovascular Safety and All-Cause Mortality of Methoxy Polyethylene Glycol-Epoetin Beta and Other Erythropoiesis-Stimulating Agents in Anemia of CKD: A Randomized Noninferiority Trial. Clin J Am Soc Nephrol. 2019 Dec 6;14(12):1701-1710. doi: 10.2215/CJN.01380219. Epub 2019 Aug 16. PMID 31420350

RESULTS

PARTICIPANT FLOW:
Groups:
- Erythropoiesis Stimulating Agents (ESA): Participants received reference ESA according to approved label. No biosimilar ESAs were accepted in the study. The approved reference ESA compounds in the study were darbepoetin alfa, epoetin alfa and epoetin beta.
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants not currently being treated with an ESA received 0.6 micrograms per kilogram (mcg/kg) methoxy polyethylene glycol-epoetin beta intravenously (iv) or subcutaneously (sc) once every 2 weeks for correction of renal anemia (target hemoglobin [Hb] 10-12 grams per deciliter [g/dL]). Participants currently treated with an ESA received a starting dose of 120, 200 or 360 mcg/kg methoxy polyethylene glycol-epoetin beta iv or sc once monthly based on the calculated weekly ESA dose prior to the switch for maintenance of anemia treatment. Once corrected and in participants currently being treated with an ESA, methoxy polyethylene glycol-epoetin beta was administered once monthly.
Period: Overall Study
Arm/Group | Erythropoiesis Stimulating Agents (ESA) | Methoxy Polyethylene Glycol-Epoetin Beta
Started (Randomized with informed consent) | 1413 | 1412
Received Study Treatment | 1409 | 1409
Completed | 312 | 303
Not Completed | 1101 | 1109
Not completed — Renal Transplant | 254 | 263
Not completed — Adverse Event / Intercurrent Illness | 40 | 48
Not completed — Withdrew Consent | 68 | 69
Not completed — Refused Treatment / Did not Cooperate | 26 | 32
Not completed — Failure to Return | 22 | 8
Not completed — Insufficient Therapeutic Response | 1 | 18
Not completed — Reason Not Specified | 159 | 126
Not completed — Death | 531 | 545

BASELINE CHARACTERISTICS:
Population: The intention-to treat (ITT) population consisted of all participants randomized with the appropriate signed consent documentation.
Groups:
- Erythropoiesis Stimulating Agents: Participants received reference ESA according to approved label. No biosimilar ESAs were accepted in the study. The approved reference ESA compounds in the study were darbepoetin alfa, epoetin alfa and epoetin beta.
- Total: Total of all reporting groups
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta | Total
Number analyzed (Participants) | 1413 | 1412 | 2825
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.8) | 62.2 (15.0) | 62.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 581 | 605 | 1186
  Male | 832 | 807 | 1639
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1221 | 1218 | 2439
  Asian | 111 | 119 | 230
  Black or African American | 40 | 37 | 77
  Other | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Time to Composite of All-Cause Mortality and Non-Fatal Cardiovascular Events (Myocardial Infarction, Stroke) Defined as Time Between First Dose of Study Medication and Date of Death or Non-Fatal Cardiovascular Events, Whichever Occurred First
Time Frame: Baseline up to approximately 8.5 years
Population: The safety population included all participants randomized (with the appropriate signed consent documentation), who received at least one dose of the trial medication and had at least one post-dose safety assessment. Data are reported for participants with an event.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
years | 5.1 [4.8 to 5.6] | 5.1 [4.7 to 5.4]
Statistical Analysis 1: Comparison: Erythropoiesis Stimulating Agents vs Methoxy Polyethylene Glycol-Epoetin Beta; Test type: Non-Inferiority — The critical alpha level for the non-inferiority test was 0.025; p = 0.0039, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.93 to 1.15] — The pre-specified upper non-inferiority limit was 95% CI <1.20

2. Secondary Outcome: Time to All-Cause Mortality
Time Frame: Baseline up to approximately 8.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
years | 6.1 [5.6 to 6.5] | 5.9 [5.5 to 6.5]
Statistical Analysis 1: Comparison: Erythropoiesis Stimulating Agents vs Methoxy Polyethylene Glycol-Epoetin Beta; Test type: Non-Inferiority — The critical alpha level for the non-inferiority test was 0.025; p = 0.0166, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.94 to 1.19]

3. Secondary Outcome: Time to Non-Fatal and Fatal Myocardial Infarction
Time Frame: Baseline up to approximately 8.5 years
Population: The safety population included all participants randomized (with the appropriate signed consent documentation), who received at least one dose of the trial medication and had at least one post-dose safety assessment. Analysis was performed on data for participants with an event.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
years | NA [NA to NA] — The median time to event was not reached. | NA [NA to NA] — The median time to event was not reached.
Statistical Analysis 1: Comparison: Erythropoiesis Stimulating Agents vs Methoxy Polyethylene Glycol-Epoetin Beta; Test type: Non-Inferiority — The critical alpha level for the non-inferiority test was 0.025; p = 0.0219, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.76 to 1.19]

4. Secondary Outcome: Time to Non-Fatal and Fatal Stroke
Time Frame: Baseline up to approximately 8.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
years | NA [NA to NA] — The median time to event was not reached. | NA [NA to NA] — The median time to event was not reached.
Statistical Analysis 1: Comparison: Erythropoiesis Stimulating Agents vs Methoxy Polyethylene Glycol-Epoetin Beta; Test type: Non-Inferiority — The critical alpha level for the non-inferiority test was 0.025; p = 0.0459, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.70 to 1.25]

5. Secondary Outcome: Time to Non-Fatal Cardiovascular Events (Myocardial Infarction or Stroke, Whichever Occurred First)
Time Frame: Baseline up to approximately 8.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
years | NA [NA to NA] — The median time to event was not reached. | NA [NA to NA] — The median time to event was not reached.
Statistical Analysis 1: Comparison: Erythropoiesis Stimulating Agents vs Methoxy Polyethylene Glycol-Epoetin Beta; Test type: Non-Inferiority — The critical alpha level for the non-inferiority test was 0.025; p = 0.0048, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.12]

6. Secondary Outcome: Percentage of Participants With Anti-Erythropoietin Antibody-Mediated Pure Red Cell Aplasia (PRCA)
Time Frame: Baseline up to approximately 8.5 years
Population: The safety population included all participants randomized (with the appropriate signed consent documentation), who received at least one dose of the trial medication and had at least one post-dose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Gastrointestinal Bleeding
Time Frame: Baseline up to approximately 8.5 years
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
percentage of participants | 11.1 | 11.7

8. Secondary Outcome: Percentage of Participants With Thromboembolic Events
Time Frame: Baseline up to approximately 8.5 years
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 1409 | 1409
percentage of participants | 34.5 | 32.8

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 8.5 years
Arm/Group | Erythropoiesis Stimulating Agents | Methoxy Polyethylene Glycol-Epoetin Beta
All-Cause Mortality (participants affected / at risk) | 557/1409 | 558/1409
Serious Adverse Events (participants affected / at risk) | 1123/1409 | 1097/1409
Other Adverse Events (participants affected / at risk) | 1171/1409 | 1177/1409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoiesis Stimulating Agents (N=1409) | Methoxy Polyethylene Glycol-Epoetin Beta (N=1409)
Pneumonia (Infections and infestations) | 163 | 180
Sepsis (Infections and infestations) | 85 | 69
Peritonitis (Infections and infestations) | 46 | 47
Septic shock (Infections and infestations) | 49 | 36
Gastroenteritis (Infections and infestations) | 27 | 39
Urinary tract infection (Infections and infestations) | 33 | 31
Device related sepsis (Infections and infestations) | 30 | 21
Lower respiratory tract infection (Infections and infestations) | 28 | 21
Cellulitis (Infections and infestations) | 25 | 22
Device related infection (Infections and infestations) | 28 | 19
Bronchitis (Infections and infestations) | 24 | 20
Gangrene (Infections and infestations) | 20 | 22
Respiratory tract infection (Infections and infestations) | 23 | 16
Staphylococcal sepsis (Infections and infestations) | 18 | 14
Urosepsis (Infections and infestations) | 11 | 19
Bacteraemia (Infections and infestations) | 14 | 10
Arteriovenous fistula site infection (Infections and infestations) | 14 | 9
Infection (Infections and infestations) | 7 | 15
Upper respiratory tract infection (Infections and infestations) | 10 | 10
Diabetic foot infection (Infections and infestations) | 9 | 10
Diverticulitis (Infections and infestations) | 13 | 5
Erysipelas (Infections and infestations) | 8 | 10
Endocarditis (Infections and infestations) | 10 | 7
Catheter site infection (Infections and infestations) | 10 | 4
Postoperative wound infection (Infections and infestations) | 10 | 4
Pyelonephritis (Infections and infestations) | 7 | 5
Staphylococcal bacteraemia (Infections and infestations) | 9 | 3
Arteriovenous graft site infection (Infections and infestations) | 7 | 4
Arthritis bacterial (Infections and infestations) | 8 | 3
Infected skin ulcer (Infections and infestations) | 8 | 3
Lung infection (Infections and infestations) | 8 | 3
Viral infection (Infections and infestations) | 3 | 8
Pyelonephritis acute (Infections and infestations) | 5 | 5
Wound infection (Infections and infestations) | 4 | 6
Escherichia sepsis (Infections and infestations) | 4 | 5
Localised infection (Infections and infestations) | 4 | 5
Pneumonia bacterial (Infections and infestations) | 4 | 5
Pulmonary sepsis (Infections and infestations) | 7 | 2
Staphylococcal infection (Infections and infestations) | 1 | 8
Influenza (Infections and infestations) | 5 | 3
Osteomyelitis (Infections and infestations) | 3 | 5
Peritonitis bacterial (Infections and infestations) | 3 | 5
Clostridium difficile colitis (Infections and infestations) | 4 | 3
Herpes zoster (Infections and infestations) | 3 | 4
Necrotising fasciitis (Infections and infestations) | 4 | 3
Renal cyst infection (Infections and infestations) | 3 | 4
Appendicitis (Infections and infestations) | 5 | 1
Bacterial sepsis (Infections and infestations) | 5 | 1
Cystitis (Infections and infestations) | 4 | 2
Diabetic gangrene (Infections and infestations) | 1 | 5
Enterococcal sepsis (Infections and infestations) | 2 | 4
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 3
Abdominal abscess (Infections and infestations) | 4 | 1
Abscess limb (Infections and infestations) | 3 | 2
Anal abscess (Infections and infestations) | 4 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 2 | 3
Infectious colitis (Infections and infestations) | 2 | 3
Infectious pleural effusion (Infections and infestations) | 3 | 2
Pseudomonal sepsis (Infections and infestations) | 1 | 4
Soft tissue infection (Infections and infestations) | 3 | 2
Abscess (Infections and infestations) | 3 | 1
Biliary sepsis (Infections and infestations) | 2 | 2
Fungal peritonitis (Infections and infestations) | 0 | 4
Gastroenteritis viral (Infections and infestations) | 3 | 1
Graft infection (Infections and infestations) | 0 | 4
H1N1 influenza (Infections and infestations) | 3 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 | 2
Ophthalmic herpes zoster (Infections and infestations) | 2 | 2
Pseudomembranous colitis (Infections and infestations) | 3 | 1
Pyelonephritis chronic (Infections and infestations) | 2 | 2
Acute sinusitis (Infections and infestations) | 3 | 0
Cellulitis gangrenous (Infections and infestations) | 2 | 1
Cholangitis infective (Infections and infestations) | 2 | 1
Cholecystitis infective (Infections and infestations) | 0 | 3
Gastroenteritis clostridial (Infections and infestations) | 2 | 1
Intervertebral discitis (Infections and infestations) | 1 | 2
Pneumonia staphylococcal (Infections and infestations) | 3 | 0
Post procedural infection (Infections and infestations) | 3 | 0
Post procedural sepsis (Infections and infestations) | 1 | 2
Pyonephrosis (Infections and infestations) | 2 | 1
Septic necrosis (Infections and infestations) | 2 | 1
Sialoadenitis (Infections and infestations) | 1 | 2
Streptococcal sepsis (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 2 | 1
Tonsillitis (Infections and infestations) | 2 | 1
Wound sepsis (Infections and infestations) | 2 | 1
Abdominal sepsis (Infections and infestations) | 2 | 0
Appendicitis perforated (Infections and infestations) | 1 | 1
Arteriosclerotic gangrene (Infections and infestations) | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 2
Empyema (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 2
Endocarditis staphylococcal (Infections and infestations) | 1 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 1
Epididymitis (Infections and infestations) | 0 | 2
Epiglottitis (Infections and infestations) | 1 | 1
Fungal oesophagitis (Infections and infestations) | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 1
Haemophilus infection (Infections and infestations) | 0 | 2
Joint tuberculosis (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 2 | 0
Listeriosis (Infections and infestations) | 0 | 2
Lymph node tuberculosis (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 1
Proteus infection (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Renal graft infection (Infections and infestations) | 0 | 2
Retroperitoneal abscess (Infections and infestations) | 2 | 0
Septic arthritis staphylococcal (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1
Skin bacterial infection (Infections and infestations) | 1 | 1
Staphylococcal skin infection (Infections and infestations) | 2 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Systemic candida (Infections and infestations) | 2 | 0
Tuberculosis (Infections and infestations) | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 1
Bacterial colitis (Infections and infestations) | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Cat scratch disease (Infections and infestations) | 1 | 0
Catheter site abscess (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Chronic tonsillitis (Infections and infestations) | 1 | 0
Citrobacter sepsis (Infections and infestations) | 1 | 0
Colon gangrene (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Corneal abscess (Infections and infestations) | 1 | 0
Corynebacterium sepsis (Infections and infestations) | 1 | 0
Cystitis bacterial (Infections and infestations) | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 0 | 1
Herpes sepsis (Infections and infestations) | 0 | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0
Infected bunion (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 1 | 0
Infective gastroduodenitis (Infections and infestations) | 0 | 1
Injection site infection (Infections and infestations) | 1 | 0
Intestinal fistula infection (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Listeria encephalitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Mesenteric abscess (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Mycetoma mycotic (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Perihepatic abscess (Infections and infestations) | 0 | 1
Periodontal destruction (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Pyomyositis (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 0 | 1
Seminal vesicle abscess (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Subacute endocarditis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1
Urethral abscess (Infections and infestations) | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 74 | 63
Atrial fibrillation (Cardiac disorders) | 57 | 49
Myocardial infarction (Cardiac disorders) | 50 | 54
Cardiac arrest (Cardiac disorders) | 44 | 55
Angina pectoris (Cardiac disorders) | 37 | 35
Cardiac failure (Cardiac disorders) | 34 | 25
Acute coronary syndrome (Cardiac disorders) | 25 | 29
Cardiac failure congestive (Cardiac disorders) | 24 | 20
Coronary artery disease (Cardiac disorders) | 24 | 20
Angina unstable (Cardiac disorders) | 16 | 24
Myocardial ischaemia (Cardiac disorders) | 21 | 17
Bradycardia (Cardiac disorders) | 20 | 8
Cardio-respiratory arrest (Cardiac disorders) | 12 | 10
Aortic valve stenosis (Cardiac disorders) | 8 | 8
Atrioventricular block complete (Cardiac disorders) | 7 | 9
Coronary artery stenosis (Cardiac disorders) | 7 | 9
Cardiogenic shock (Cardiac disorders) | 9 | 5
Atrial flutter (Cardiac disorders) | 9 | 4
Cardiac failure acute (Cardiac disorders) | 4 | 9
Cardiopulmonary failure (Cardiac disorders) | 3 | 8
Ventricular fibrillation (Cardiac disorders) | 3 | 7
Arrhythmia (Cardiac disorders) | 7 | 2
Left ventricular failure (Cardiac disorders) | 5 | 4
Cardiac failure chronic (Cardiac disorders) | 5 | 2
Atrioventricular block (Cardiac disorders) | 4 | 2
Cardiomyopathy (Cardiac disorders) | 5 | 1
Sinus node dysfunction (Cardiac disorders) | 4 | 2
Ventricular tachycardia (Cardiac disorders) | 2 | 3
Aortic valve disease (Cardiac disorders) | 2 | 2
Atrial tachycardia (Cardiac disorders) | 4 | 0
Atrioventricular block second degree (Cardiac disorders) | 3 | 1
Pericardial effusion (Cardiac disorders) | 2 | 2
Pericarditis (Cardiac disorders) | 2 | 2
Sinus bradycardia (Cardiac disorders) | 2 | 2
Acute left ventricular failure (Cardiac disorders) | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 0
Atrial thrombosis (Cardiac disorders) | 3 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 2
Coronary artery thrombosis (Cardiac disorders) | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 2 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 2
Aortic valve disease mixed (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 2
Pericarditis uraemic (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Chordae tendinae rupture (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Diabetic cardiomyopathy (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1
Heart valve stenosis (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Paroxysmal atrioventricular block (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular dyssynchrony (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 110 | 77
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 57 | 47
Femur fracture (Injury, poisoning and procedural complications) | 23 | 26
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 16 | 23
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 13 | 23
Femoral neck fracture (Injury, poisoning and procedural complications) | 19 | 14
Procedural hypotension (Injury, poisoning and procedural complications) | 13 | 16
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 15 | 6
Subdural haematoma (Injury, poisoning and procedural complications) | 8 | 12
Hip fracture (Injury, poisoning and procedural complications) | 8 | 11
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 11 | 7
Rib fracture (Injury, poisoning and procedural complications) | 8 | 9
Head injury (Injury, poisoning and procedural complications) | 9 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 7 | 7
Fall (Injury, poisoning and procedural complications) | 8 | 5
Multiple fractures (Injury, poisoning and procedural complications) | 5 | 8
Overdose (Injury, poisoning and procedural complications) | 6 | 5
Pelvic fracture (Injury, poisoning and procedural complications) | 8 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 7
Limb injury (Injury, poisoning and procedural complications) | 5 | 4
Radius fracture (Injury, poisoning and procedural complications) | 5 | 4
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 4 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 6 | 2
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 3 | 5
Lower limb fracture (Injury, poisoning and procedural complications) | 4 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 6
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 4
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 | 3
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 5
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 5 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 4
Anaemia postoperative (Injury, poisoning and procedural complications) | 4 | 1
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 4 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 4
Forearm fracture (Injury, poisoning and procedural complications) | 3 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 4 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 4 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 2
Concussion (Injury, poisoning and procedural complications) | 2 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 2
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 3
Muscle rupture (Injury, poisoning and procedural complications) | 2 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 2
Wound necrosis (Injury, poisoning and procedural complications) | 2 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 2 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 1
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 2
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 2
Procedural complication (Injury, poisoning and procedural complications) | 1 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 1
Shunt aneurysm (Injury, poisoning and procedural complications) | 2 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 1
Skin wound (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 1
Device deployment issue (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 1
Extensive interdialytic weight gain (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Haemodialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Stomal hernia (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic coma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 23 | 24
Abdominal pain (Gastrointestinal disorders) | 16 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 18
Large intestine polyp (Gastrointestinal disorders) | 10 | 9
Rectal haemorrhage (Gastrointestinal disorders) | 8 | 10
Gastritis (Gastrointestinal disorders) | 11 | 5
Constipation (Gastrointestinal disorders) | 8 | 7
Gastric ulcer (Gastrointestinal disorders) | 5 | 10
Inguinal hernia (Gastrointestinal disorders) | 7 | 8
Colitis ischaemic (Gastrointestinal disorders) | 7 | 7
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 8 | 6
Intestinal ischaemia (Gastrointestinal disorders) | 9 | 5
Intestinal obstruction (Gastrointestinal disorders) | 9 | 5
Melaena (Gastrointestinal disorders) | 7 | 7
Colitis (Gastrointestinal disorders) | 8 | 5
Pancreatitis acute (Gastrointestinal disorders) | 9 | 3
Pancreatitis (Gastrointestinal disorders) | 5 | 6
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 6 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3
Gastritis erosive (Gastrointestinal disorders) | 3 | 6
Gastritis haemorrhagic (Gastrointestinal disorders) | 6 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 7
Umbilical hernia (Gastrointestinal disorders) | 7 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 5
Diverticulum (Gastrointestinal disorders) | 5 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 5
Enteritis (Gastrointestinal disorders) | 5 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 4 | 3
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 3 | 3
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 3 | 3
Haematemesis (Gastrointestinal disorders) | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 3
Intestinal infarction (Gastrointestinal disorders) | 4 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 3 | 2
Chronic gastritis (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 4
Large intestine perforation (Gastrointestinal disorders) | 1 | 3
Subileus (Gastrointestinal disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 2
Acute abdomen (Gastrointestinal disorders) | 2 | 1
Anal fistula (Gastrointestinal disorders) | 2 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 1
Encapsulating peritoneal sclerosis (Gastrointestinal disorders) | 2 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 2 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal angiectasia (Gastrointestinal disorders) | 2 | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 3 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 3
Ileus (Gastrointestinal disorders) | 1 | 2
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 3
Necrotising colitis (Gastrointestinal disorders) | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal prolapse (Gastrointestinal disorders) | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis erosive (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 2
Erosive duodenitis (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 2 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 0
Peritoneal perforation (Gastrointestinal disorders) | 2 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal stenosis (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Anorectal varices (Gastrointestinal disorders) | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Diabetic gastropathy (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum oesophageal (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal varices (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Ischaemic enteritis (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 31 | 31
Peripheral arterial occlusive disease (Vascular disorders) | 24 | 24
Hypertension (Vascular disorders) | 24 | 23
Hypotension (Vascular disorders) | 18 | 16
Extremity necrosis (Vascular disorders) | 13 | 10
Hypertensive crisis (Vascular disorders) | 8 | 13
Peripheral artery stenosis (Vascular disorders) | 8 | 12
Peripheral vascular disorder (Vascular disorders) | 11 | 9
Aortic stenosis (Vascular disorders) | 11 | 5
Deep vein thrombosis (Vascular disorders) | 9 | 7
Orthostatic hypotension (Vascular disorders) | 7 | 8
Haematoma (Vascular disorders) | 5 | 9
Shock haemorrhagic (Vascular disorders) | 6 | 5
Aortic aneurysm (Vascular disorders) | 5 | 5
Steal syndrome (Vascular disorders) | 2 | 8
Dry gangrene (Vascular disorders) | 4 | 5
Intermittent claudication (Vascular disorders) | 3 | 5
Peripheral artery occlusion (Vascular disorders) | 5 | 3
Venous stenosis (Vascular disorders) | 4 | 4
Circulatory collapse (Vascular disorders) | 3 | 4
Aortic aneurysm rupture (Vascular disorders) | 2 | 4
Brachiocephalic vein stenosis (Vascular disorders) | 3 | 3
Peripheral artery thrombosis (Vascular disorders) | 2 | 4
Angiopathy (Vascular disorders) | 4 | 1
Arterial disorder (Vascular disorders) | 3 | 2
Granulomatosis with polyangiitis (Vascular disorders) | 3 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 3
Vena cava thrombosis (Vascular disorders) | 3 | 1
Venous thrombosis limb (Vascular disorders) | 3 | 1
Arterial occlusive disease (Vascular disorders) | 2 | 1
Shock (Vascular disorders) | 1 | 2
Superior vena cava syndrome (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 0 | 3
Angiodysplasia (Vascular disorders) | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 1
Arterial haemorrhage (Vascular disorders) | 1 | 1
Arterial rupture (Vascular disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 1 | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 2 | 0
Diabetic macroangiopathy (Vascular disorders) | 0 | 2
Diabetic vascular disorder (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 1
Leriche syndrome (Vascular disorders) | 0 | 2
Peripheral embolism (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 1
Subclavian vein stenosis (Vascular disorders) | 0 | 2
Thrombophlebitis (Vascular disorders) | 1 | 1
Vascular calcification (Vascular disorders) | 0 | 2
Venous thrombosis (Vascular disorders) | 0 | 2
Aneurysm (Vascular disorders) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Femoral artery dissection (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1
Ischaemic limb pain (Vascular disorders) | 0 | 1
Lymphatic fistula (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Lymphostasis (Vascular disorders) | 0 | 1
Microangiopathy (Vascular disorders) | 1 | 0
Microscopic polyangiitis (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Vasculitis necrotising (Vascular disorders) | 1 | 0
Venous aneurysm (Vascular disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 28 | 21
Cerebrovascular accident (Nervous system disorders) | 23 | 24
Transient ischaemic attack (Nervous system disorders) | 17 | 30
Syncope (Nervous system disorders) | 22 | 15
Cerebral haemorrhage (Nervous system disorders) | 7 | 8
Seizure (Nervous system disorders) | 10 | 5
Cerebral infarction (Nervous system disorders) | 4 | 9
Dizziness (Nervous system disorders) | 4 | 9
Carpal tunnel syndrome (Nervous system disorders) | 7 | 3
Cerebral ischaemia (Nervous system disorders) | 4 | 6
Haemorrhagic stroke (Nervous system disorders) | 7 | 3
Haemorrhage intracranial (Nervous system disorders) | 5 | 4
Dementia (Nervous system disorders) | 3 | 5
Sciatica (Nervous system disorders) | 5 | 3
Epilepsy (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 3 | 3
Hepatic encephalopathy (Nervous system disorders) | 3 | 3
Carotid artery stenosis (Nervous system disorders) | 2 | 3
Vascular dementia (Nervous system disorders) | 2 | 3
Cerebrovascular disorder (Nervous system disorders) | 2 | 2
Presyncope (Nervous system disorders) | 3 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 3
Altered state of consciousness (Nervous system disorders) | 2 | 1
Cerebral haematoma (Nervous system disorders) | 3 | 0
Dementia Alzheimer's type (Nervous system disorders) | 3 | 0
Facial paralysis (Nervous system disorders) | 1 | 2
Hypertensive encephalopathy (Nervous system disorders) | 1 | 2
Stupor (Nervous system disorders) | 1 | 2
Aphasia (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 2
Brain stem infarction (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 2 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 1
Intraventricular haemorrhage (Nervous system disorders) | 2 | 0
Lacunar infarction (Nervous system disorders) | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 2
Polyneuropathy (Nervous system disorders) | 1 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 2
Balance disorder (Nervous system disorders) | 1 | 0
Brain hypoxia (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral ataxia (Nervous system disorders) | 1 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Demyelination (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Diabetic mononeuropathy (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Essential tremor (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypocalcaemic seizure (Nervous system disorders) | 1 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic neuropathy (Nervous system disorders) | 0 | 1
IVth nerve paresis (Nervous system disorders) | 0 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Noninfective encephalitis (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Retrograde amnesia (Nervous system disorders) | 0 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Wallerian degeneration (Nervous system disorders) | 0 | 1
Death (General disorders) | 33 | 39
Sudden death (General disorders) | 26 | 44
Pyrexia (General disorders) | 30 | 26
General physical health deterioration (General disorders) | 16 | 12
Chest pain (General disorders) | 13 | 10
Catheter site haemorrhage (General disorders) | 7 | 7
Non-cardiac chest pain (General disorders) | 11 | 3
Asthenia (General disorders) | 7 | 2
Inflammation (General disorders) | 4 | 5
Multiple organ dysfunction syndrome (General disorders) | 6 | 3
Complication associated with device (General disorders) | 3 | 5
Sudden cardiac death (General disorders) | 4 | 3
Hyperthermia (General disorders) | 5 | 1
Adverse drug reaction (General disorders) | 0 | 4
Device related thrombosis (General disorders) | 1 | 3
Hyperpyrexia (General disorders) | 1 | 3
Malaise (General disorders) | 3 | 1
Oedema due to renal disease (General disorders) | 2 | 2
Fatigue (General disorders) | 2 | 1
Hernia (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 2
Swelling (General disorders) | 3 | 0
Catheter site inflammation (General disorders) | 1 | 1
Chest discomfort (General disorders) | 2 | 0
Gait disturbance (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 1
Strangulated hernia (General disorders) | 2 | 0
Systemic inflammatory response syndrome (General disorders) | 2 | 0
Accidental death (General disorders) | 1 | 0
Discomfort (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Dysplasia (General disorders) | 1 | 0
Heteroplasia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site extravasation (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Injection site extravasation (General disorders) | 0 | 1
Injection site scab (General disorders) | 0 | 1
Medical device pain (General disorders) | 0 | 1
Mucosal ulceration (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Oedema due to cardiac disease (General disorders) | 1 | 0
Pseudocyst (General disorders) | 0 | 1
Stent-graft endoleak (General disorders) | 1 | 0
Surgical failure (General disorders) | 1 | 0
Treatment failure (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1
Vascular stent thrombosis (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22 | 22
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 16
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mendelson's syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of epididymis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Connective tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extranodal marginal zone B-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 44 | 43
Hyperkalaemia (Metabolism and nutrition disorders) | 18 | 32
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 17
Cachexia (Metabolism and nutrition disorders) | 9 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 7
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 6
Malnutrition (Metabolism and nutrition disorders) | 4 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 4
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 4
Diabetic complication (Metabolism and nutrition disorders) | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Mitochondrial cytopathy (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 31 | 26
Renal impairment (Renal and urinary disorders) | 20 | 18
Haematuria (Renal and urinary disorders) | 7 | 8
Chronic kidney disease (Renal and urinary disorders) | 7 | 4
Azotaemia (Renal and urinary disorders) | 4 | 6
Acute kidney injury (Renal and urinary disorders) | 6 | 3
Nephrolithiasis (Renal and urinary disorders) | 2 | 4
Renal cyst haemorrhage (Renal and urinary disorders) | 2 | 3
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Renal failure (Renal and urinary disorders) | 1 | 3
Renal colic (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 3 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 1
Bladder tamponade (Renal and urinary disorders) | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Kidney enlargement (Renal and urinary disorders) | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 1
Malnutrition-inflammation-atherosclerosis syndrome (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal ischaemia (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 16
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 4
Osteitis (Musculoskeletal and connective tissue disorders) | 2 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Collagen disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
High turnover osteopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 10 | 12
Cholecystitis acute (Hepatobiliary disorders) | 13 | 7
Cholelithiasis (Hepatobiliary disorders) | 7 | 8
Cholangitis (Hepatobiliary disorders) | 5 | 5
Jaundice cholestatic (Hepatobiliary disorders) | 4 | 1
Bile duct stone (Hepatobiliary disorders) | 3 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 2
Cholestasis (Hepatobiliary disorders) | 2 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Haemobilia (Hepatobiliary disorders) | 1 | 0
Hepatic artery stenosis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 17 | 17
Diabetic foot (Skin and subcutaneous tissue disorders) | 13 | 11
Skin necrosis (Skin and subcutaneous tissue disorders) | 3 | 3
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 2
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 22 | 25
Haemolysis (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 2
Anaemia of malignant disease (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 19 | 23
Hyperparathyroidism tertiary (Endocrine disorders) | 4 | 4
Adrenal insufficiency (Endocrine disorders) | 3 | 2
Hyperparathyroidism (Endocrine disorders) | 3 | 1
Goitre (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 3
Basedow's disease (Endocrine disorders) | 1 | 1
Parathyroid hyperplasia (Endocrine disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 14 | 10
Delirium (Psychiatric disorders) | 3 | 3
Completed suicide (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 2 | 2
Hallucination (Psychiatric disorders) | 1 | 2
Sopor (Psychiatric disorders) | 1 | 2
Adjustment disorder (Psychiatric disorders) | 1 | 1
Mania (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 2 | 0
Organic brain syndrome (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 2 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Device malfunction (Product Issues) | 7 | 8
Thrombosis in device (Product Issues) | 6 | 9
Device dislocation (Product Issues) | 4 | 1
Device loosening (Product Issues) | 3 | 1
Device breakage (Product Issues) | 1 | 0
Device damage (Product Issues) | 0 | 1
Device extrusion (Product Issues) | 1 | 0
Device failure (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Cataract (Eye disorders) | 9 | 10
Vitreous haemorrhage (Eye disorders) | 4 | 2
Glaucoma (Eye disorders) | 2 | 3
Diabetic retinopathy (Eye disorders) | 1 | 3
Retinal artery occlusion (Eye disorders) | 1 | 1
Cataract diabetic (Eye disorders) | 1 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 1
Ocular vasculitis (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 1 | 0
Retinal neovascularisation (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Vitreous haematoma (Eye disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Prostatitis (Reproductive system and breast disorders) | 1 | 3
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
Breast mass (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Hysterocele (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 4 | 2
Hypersensitivity (Immune system disorders) | 4 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 2 | 1
Kidney transplant rejection (Immune system disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Graft versus host disease (Immune system disorders) | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1
Pancreas transplant rejection (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 3
International normalised ratio increased (Investigations) | 0 | 2
Coagulation time prolonged (Investigations) | 0 | 1
Investigation abnormal (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 2
Hydrocele (Congenital, familial and genetic disorders) | 0 | 2
Congenital bladder anomaly (Congenital, familial and genetic disorders) | 0 | 1
Nonketotic hyperglycinaemia (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Oral surgery (Surgical and medical procedures) | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoiesis Stimulating Agents (N=1409) | Methoxy Polyethylene Glycol-Epoetin Beta (N=1409)
Nasopharyngitis (Infections and infestations) | 171 | 187
Bronchitis (Infections and infestations) | 195 | 188
Urinary tract infection (Infections and infestations) | 193 | 200
Upper respiratory tract infection (Infections and infestations) | 153 | 132
Gastroenteritis (Infections and infestations) | 93 | 101
Pneumonia (Infections and infestations) | 101 | 79
Respiratory tract infection (Infections and infestations) | 76 | 70
Lower respiratory tract infection (Infections and infestations) | 55 | 74
Influenza (Infections and infestations) | 83 | 72
Diarrhoea (Gastrointestinal disorders) | 269 | 273
Constipation (Gastrointestinal disorders) | 173 | 142
Vomiting (Gastrointestinal disorders) | 146 | 121
Nausea (Gastrointestinal disorders) | 99 | 104
Abdominal pain (Gastrointestinal disorders) | 88 | 102
Abdominal pain upper (Gastrointestinal disorders) | 70 | 82
Dyspepsia (Gastrointestinal disorders) | 78 | 59
Muscle spasms (Musculoskeletal and connective tissue disorders) | 211 | 199
Back pain (Musculoskeletal and connective tissue disorders) | 158 | 119
Pain in extremity (Musculoskeletal and connective tissue disorders) | 133 | 124
Arthralgia (Musculoskeletal and connective tissue disorders) | 110 | 125
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 105 | 86
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 79 | 72
Hypertension (Vascular disorders) | 432 | 455
Hypotension (Vascular disorders) | 143 | 124
Procedural hypotension (Injury, poisoning and procedural complications) | 225 | 223
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 171 | 158
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 87 | 86
Hyperkalaemia (Metabolism and nutrition disorders) | 140 | 122
Hyperphosphataemia (Metabolism and nutrition disorders) | 142 | 136
Fluid overload (Metabolism and nutrition disorders) | 130 | 115
Cough (Respiratory, thoracic and mediastinal disorders) | 194 | 162
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 109 | 109
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 72 | 50
Pyrexia (General disorders) | 96 | 92
Oedema due to renal disease (General disorders) | 79 | 78
Asthenia (General disorders) | 59 | 85
Oedema peripheral (General disorders) | 73 | 61
Headache (Nervous system disorders) | 127 | 141
Dizziness (Nervous system disorders) | 78 | 81
Insomnia (Psychiatric disorders) | 116 | 104
Depression (Psychiatric disorders) | 65 | 75
Anaemia (Blood and lymphatic system disorders) | 143 | 174
Hyperparathyroidism secondary (Endocrine disorders) | 149 | 148
Atrial fibrillation (Cardiac disorders) | 123 | 111
Pruritus (Skin and subcutaneous tissue disorders) | 118 | 114
Cataract (Eye disorders) | 72 | 76

LIMITATIONS AND CAVEATS:
The study was designed and powered to formally test only the primary composite outcome measure only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT00773513/Prot_SAP_000.pdf